CLINICAL TRIAL: NCT06550648
Title: Evaluation of the Role of Epstein-Bar Virus in Patients With Pulmonary Arterial Hypertension
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Yasser Mohammed Elhalafawy, Dr, Cairo University
Other Study IDs: MD-110-2023
Record Dates: First submitted 2024-07-19; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 5cc of Serum Blood Sample for assessment of EBV Immunoglobulins (IgG and IgM) and PCR .
  Routine RHC by disposable balloon tipped Swan Ganz catheter is performed for diagnosis. After the procedure the tip of the catheter (including the balloon) will be separated and put in a sterile cup then transferred to the clinical pathology lab within 20 mins for isolation of endothelial cell and culturing the virus if present.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Idiopathic Pulmonary Arterial Hypertension: Patients with Idiopathic PAH excluding all other causes Right Heart Catheterization will be done as routine as well as blood samples for IgG and IgM and EBV PCR
  Interventions: Procedure: Right Heart Catheterization (Swan Ganz Catheter)
- Pulmonary Arterial Hypertension associated with Connective Tissue Disease: Proved CTD Right Heart Catheterization will be done as routine as well as blood samples for IgG and IgM and EBV PCR
  Interventions: Procedure: Right Heart Catheterization (Swan Ganz Catheter)
- Control group ( Normal Individuals ): Healthy Individuals ( only Blood samples withdrawn)

INTERVENTIONS:
Procedure: Right Heart Catheterization (Swan Ganz Catheter) — Swan Ganz Catheter only for PAH patients, Using the swan ganz and pressure transducer
  Groups: Idiopathic Pulmonary Arterial Hypertension; Pulmonary Arterial Hypertension associated with Connective Tissue Disease

SUMMARY:
Evaluate the role of Epstein-Barr virus infection in PAH (Idiopathic and connective tissue disease).

This by obtaining a blood sample from the PAH patients undergoing right heart cathetrization as well as obtaining the endothelial cells from the balloon tipped catheters and extracting the EBV virus to detect its presence.

IgG, IgM and PCR for EBV tests will be done.

DETAILED DESCRIPTION:
About Pulmonary Hypertension Pulmonary hypertension (PH) is a pathophysiological disorder that may involve multiple clinical conditions combined with a variety of cardiovascular and respiratory diseases. It is defined by a mean pulmonary arterial pressure (mPAP) of more than 20 mmHg at rest (Humbert, M.et al., 2022).

Pulmonary arterial hypertension (PAH) is a condition characterized by vascular proliferation, leading to increased vascular resistance and right heart dysfunction. PAH may be idiopathic (Idiopathic Pulmonary Arterial Hypertension IPAH; previously known as primary pulmonary hypertension, PPH) or associated with other conditions or exposures, including connective tissue diseases, HIV infection, portal hypertension, and anorexigenic drug ingestion (Humbert, M.et al., 2022).

About Chronic active Epstein-Barr virus Chronic Active Epstein-Barr virus (CAEBV) disease is usually defined as a chronic illness lasting at least 6 months, an increased EBV level in either the tissue or the blood, and lack of evidence of a known underlying immunodeficiency. It may be associated with Burkitt lymphoma and nasopharyngeal carcinoma, Hodgkin lymphoma, peripheral T cell lymphoma, angioimmunoblastic T cell lymphoma, and extranodal NK/T cell lymphoma (Kimura et al., 2017).

CAEBV is characterized by an unusual pattern of anti-EBV antibodies and may be associated with cardiovascular abnormalities (Hashimoto et al., 2011).

Diagnosis of Epstein-Barr virus (EBV) infection is based on clinical symptoms and serological markers, including the following: immunoglobulin G (IgG) and IgM antibodies to the viral capsid antigen (VCA), heterophile antibodies, and IgG antibodies to the EBV early antigen-diffuse (EA-D) and nuclear antigen (EBNA-1)(Klutts JS. Et al., 2009).

Elevated levels of EBV DNA in the blood are more specific for CAEBV than elevated levels of EBV antibodies (Kimura H. et al., 2017).

Role of EBV in PAH The relationships between EBV and autoimmune diseases are complex and involve several mechanisms. A proposed scenario was the interrelation between genetic predisposition and EBV infection, a cross-reaction between self antigens and EBV viral proteins, the development of autoantibodies (anti-Sm or anti-Ro antibodies in SLE, anti-CCP antibodies in RA), an epitope-spreading process that can lead to the development of additional non-cross-reactive autoepitopes, and finally the clinical manifestations (Poole BD et al.,2006).

EBV has multiple impacts on host immunity and can adapt to its environment. For instance, EBV produces an IL-10-like cytokine, it can modulate IL-6 release, it induces the production of TNF-a by infected B cells, and it can inhibit apoptosis of infected B cells by the production of a Bcl-2 homolog. All these biological properties of EBV are relevant to, and can contribute to, the pathophysiology of autoimmune disorders (Toussirot É et al.,2008).

The pathophysiology of the development of PAH in CAEBV is unclear. It may be related to lymphocytic infiltration and the resultant damage to the pulmonary vascular endothelium caused by EBV infection or may occur secondary to the vascular damage caused by inflammatory reactions induced by EBV infection (Gotoh K. et al., 2008).

Another is EBV-induced high levels of inflammatory cytokines resulting in inflammatory change (Fujiwara M. et al., 2003).

ELIGIBILITY:
Inclusion Criteria:

* Group 1 PAH (Idiopathic ) Group 1 PAH ( Connective tissue disease including SLE, Systemic sclerosis and mixed connective tissue disease) Above 18 years

Exclusion Criteria:

* Other Groups of Pulmonary hypertension Patients refusing written consent or participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PAH patients (Idiopathic and connective tissue disease; inclusing SLE , systemic sclerosis and mixed connective tissue disease).
  Control group: Healthy individuals only blood samples withdrawn
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
EBV PCR and Immunoglobulins in patients with PAH test will be done | from may 2023 till july 2024
  by virus detection in both blood and endothelial cells and its immunoglobulins
The percentage of EBV-positive patients to normal control subjects | from may 2023 till july 2024
  Test results statically analyzed to corelate
The presence of EBV within the endothelial cell line in patients | from may 2023 till july 2024
  PCR of the virus in the endothelial cell culture proving the viral invasion causing the remodeling

SECONDARY OUTCOMES:
CAEBV-infected individual 's risk assessment compared to the risk assessment of those who are not infected. | from may 2023 till july 2024
  by three risk strata assessment to all patients

CONTACTS AND LOCATIONS:
Overall Officials: Hoda MM Abdel-Hamid, MD, Study Chair — Assistant Professor; Jumana H Ismail, MD, Study Chair — Lecturer; Hala G Metwally, MD, Study Chair — Professor
Locations (1):
- Cairo University- Faculty Of Medicine, Cairo, Egypt